CLINICAL TRIAL: NCT05500599
Title: Effects on Recovery of Children Undergoing Elective Surgery: Comparison of Intravenous Formulation of Fentanyl Citrate and Midazolam Administered Orally for Premedication
Brief Title: Effects on Recovery of Children of Intravenous Formulation of Fentanyl Citrate and Midazolam Orally for Premedication
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Ahmed Shehab, MD, lecturer Of Anaesthesia and Surgical intensive care, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 0305335
Record Dates: First submitted 2022-08-10; First posted 2022-08-15 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Separation Anxiety
Keywords: recovery; Anxiety; Fentanyl; midazolam; Premedication
MeSH Terms: conditions — Anxiety, Separation; Anxiety Disorders | interventions — Fentanyl; Midazolam

STUDY DESIGN:
Intervention Model Description: All children will be randomized to one of two groups of thirty patients each according to a computer-generated random numbers program in a double-blinded fashion, to receive either 0.5 mg/kg midazolam (Group M) or 10 μg/kg fentanyl (Group F) approximately 30 min before the induction of anaesthesia. All observers, as well as the children and their parents, will be blind to the study drug administered.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- midazolam (Group M) (No Intervention): receive 0.5 mg/kg midazolam orally approximately 30 min before the induction of anaesthesia
- fentanyl (Group F) (Active Comparator): receive 10 μg/kg fentanyl orally approximately 30 min before the induction of anaesthesia
  Interventions: Drug: Fentanyl Citrate

INTERVENTIONS:
Drug: Fentanyl Citrate — Intravenous Formulation of Fentanyl Citrate and Midazolam Administered Orally for Premedication
  Other Names: Midazolam
  Arms: fentanyl (Group F)

SUMMARY:
To study and compare the efficacy of intravenous formula of fentanyl citrate and midazolam administered orally for premedication in paediatric surgical patients. Primary objectives will be the effect of both premedicants on recovery. The secondary outcomes will be time of onset and level of sedation, acceptance of premedication, and adverse effects. Sixty paediatric patients of either sex, in the age group of 2-8 years, with the American Society of Anaesthesiologists (ASA) Physical status I, posted for elective Genito-urological surgeries under general anaesthesia (GA) will be studied after clearance from the Institutional Ethics Committee and after obtaining written informed consent from a parent or a legal guardian

DETAILED DESCRIPTION:
Effects on Recovery of Children Undergoing Elective Surgery: Comparison of Intravenous Formulation of Fentanyl Citrate and Midazolam Administered Orally for Premedication

Introduction Paediatric preoperative anxiety has been a concerning matter for the past decades with a high prevalence and several adverse outcomes branching into social, developmental, behavioural, and perioperative fields. The anticipation of pain, separation from family, and fear of surgery are few of the factors that trigger perioperative anxiety in children. However, the routine use of anxiolytic premedication before anaesthetic induction is debated. Furthermore, premedication may significantly affect recovery from anaesthesia.

Premedication causes sedation and reduction of anxiety during separation from parents. It also provides a calm and cooperative child for smooth induction of anaesthesia. The oral route of administration of the drugs is the most acceptable and a nontraumatic route, especially in children. The total volume of the oral premedication can be kept at 0.2 ml/kg which is far below the gastric fluid volume of 0.4 ml/kg above which the risk of aspiration increases. Lipid-soluble drugs that can be supplied as water-soluble salts provide the opportunity to use it through oral route of administration for premedication.

The salt fentanyl citrate is soluble in water. These properties suggest that fentanyl citrate can be incorporated for use as a premedicant. This lipid-soluble opioid when placed in normal conditions of the mouth is 80% nonionized, making it the only opioid suitable for transmucosal absorption. However, bioavailability depends on the fraction of the dose that is absorbed through the oral mucosa (~25%) and the fraction that is swallowed (~75%, swallowed dose is only partially bioavailable).

Midazolam, a benzodiazepine, has been routinely used orally for premedication in children scheduled for surgery. Bioavailability of oral midazolam varies from 15% to 27% in children. It has a rapid onset and short duration of action. It is reliable in achieving sedation and anxiolysis. However, search for a better alternative continues due to concerns such as bitter taste, cognitive impairment, long-term behavioural disturbances, paradoxical reactions, hiccups, and respiratory depression.

Aim: To study and compare the efficacy of intravenous formula of fentanyl citrate and midazolam administered orally for premedication in paediatric surgical patients.

Objectives: The primary objectives will be the effect of both premedicants on recovery. The secondary outcomes will be time of onset and level of sedation, acceptance of premedication, and adverse effects.

Settings and Design: This prospective, randomized, double blind study will be conducted in Alexandria Main University hospital.

Materials and Methods Sixty paediatric patients of either sex, in the age group of 2-8 years, with the American Society of Anaesthesiologists (ASA) Physical status I, posted for elective Genito-urological surgeries under general anaesthesia (GA) will be studied after clearance from the Institutional Ethics Committee and after obtaining written informed consent from a parent or a legal guardian.

Patients with known allergy to fentanyl or midazolam, intellectual and developmental disabilities, psychosomatic disorders, history of any sedative or analgesic intake, ASA physical status ≥ 2, those with upper respiratory tract infection, history of previous surgery, and being accompanied by a non-family member will not be included in the study.

All children will be randomized to one of two groups of thirty patients each according to a computer-generated random numbers program in a double-blinded fashion, to receive either 0.5 mg/kg midazolam (Group M) or 10 μg/kg fentanyl (Group F) approximately 30 min before the induction of anaesthesia. All observers, as well as the children and their parents, will be blind to the study drug administered.

Children will be fasted 4-6 h before surgery. Before administration of the premedication, the children will be taken to the preoperative anaesthetic assessment area along with their family members. An intravenous preparation of a drug (midazolam 5 mg/ml solution, or fentanyl 50 µg/ml solution) will be mixed with apple juice a to total volume not exceeding 0.3 ml/kg body weight and given orally.

The children will be separated from their family members and taken to the operating room (OR) 30 min after the administration of premedication. In the OR, electrocardiograph, non-invasive blood pressure, and pulse oximetry monitors will be attached. Inhalation induction will be performed using sevoflurane in 100 % oxygen. An intravenous line will be secured, and fentanyl 1 µg/kg will be given intravenously for analgesia, and muscle relaxation will be provided with intravenous atracurium 0.5 mg/kg. Endotracheal tube of an appropriate size will be inserted 3 min after the administration of the muscle relaxant and capnography will be connected. Regional analgesia will be applied according to type of surgery. Measures to prevent hypothermia will be performed (e.g., warming blanket, warming intravenous fluids, etc.). Anaesthesia will be maintained with sevoflurane (2-3%), oxygen and air, and supplemental doses of atracurium 0.25 mg/kg. At the end of surgery intravenous paracetamol suppository in the dose of 15 mg/kg will be used for postoperative analgesia. Inhalational agent will be switched off, and effect of muscle relaxant will be reversed with neostigmine (0.05 mg/kg) and atropine (0.01 mg/kg) given intravenously. The patient will be extubated following return of regular, rhythmic respiration when reasonably awake. Patients will be shifted to the postoperative recovery room for observation and will be given oxygen inhalation by venturi mask. Parents will be allowed to join children.

Measurements:

1. Children's anxiety will be assessed using the modified Yale Preoperative Anxiety Scale-Short Version at the preoperative holding area before receiving medication (Time 1), and in the operating room after separation from the parent (Time 2), where the children will not be accompanied by their family.

   The total score of the scale will be calculated as suggested by the authors that revised the scale. For each domain the patient's partial score will be divided by the maximum score obtainable in that domain (6 for the vocalizations domain and 4 for the remaining). The produced values for each domain are all added up and multiplied by 25. A score ranging from 22.92 to 100 will be obtained with higher values, representing higher states of anxiety. Thus, for study purposes, children with scores more than 30 will be considered as having anxiety and children with scores from 22,92 to 30 will be considered as not having experienced significant anxiety.
2. Acceptance of premedication will be assessed on a three-point scale; 1 = Accepts it/likes the taste, 2 = Accepts it/but dislikes the taste. 3 = Spits/vomits the premedication. Score of 1 or 2 will be judged as satisfactory acceptance of oral premedication.
3. Degree and onset of sedation will be assessed 15 and 30 minutes after administration of premedication by Ramsay sedation scale. Scale scored from 1 (least sedated) to 6 (most sedated).
4. Behaviour of the child on separation from parents will be rated according to a four-point scale, i.e., the parental separation anxiety scale (PSAS): A PSAS score of 1 and 2 will be considered as acceptable separation from parents. A PSAS score of 3 and 4 will be considered as non-acceptable separation from parents
5. Mask acceptance will be recorded using a four-point scale. The score of 1 and 2 will be considered as satisfactory mask acceptance. The score of 3 and 4 will be considered as satisfactory mask acceptance.
6. Assessment of recovery:

   i. Emergence time (minutes): from discontinuation of anaesthesia to opening eyes spontaneously will be recorded.

   ii. Recovery time (minutes): from discontinuation of anaesthesia to a score of 8 on the modified Aldrete score will be recorded.

   iii. The quality of recovery will be evaluated using the three objective components in the modified pain/discomfort scale, each variable scoring 0-2 points (best to worst). If the total score on the pain/discomfort scale at any evaluation point exceeded 3, the child will be regarded as suffering from postanaesthetic excitement.

7) Adverse effects: children will be observed for adverse effects if any before they left the preoperative area, and again after the surgery before they left the recovery area. Adverse effects such as hypotension, bradycardia, bradypnea or apnoea, fall in saturation, shivering, vomiting, nausea, pruritus, headache and hiccups if any will be noted for 2 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* (ASA) Physical status I,
* posted for elective Genito-urological surgeries under general anaesthesia (GA)

Exclusion Criteria:

* known allergy to fentanyl or midazolam,
* intellectual and developmental disabilities,
* psychosomatic disorders,
* history of any sedative or analgesic intake,
* ASA physical status ≥ 2,
* upper respiratory tract infection,
* history of previous surgery,
* being accompanied by a non-family member

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-08-28 (Estimated)

PRIMARY OUTCOMES:
effect of both premedicants on recovery | immediately after the surgery average 2 hours postoperative
  1. The quality of recovery will be evaluated using the three objective components in the modified pain/discomfort scale. Each variable scoring 0-2 points (best to worst). If the total score on the pain/discomfort scale at any evaluation point exceeded 3, the child will be regarded as suffering from postanaesthetic excitement.
  score 0 1 2 Crying Not crying Responding to pain Not responding to comforting Moving None Restless Thrashing Agitation Asleep/calm Mild agitation Sever agitation/Hysterical

SECONDARY OUTCOMES:
time of onset and level of sedation, | Before the surgery starts
  1. Children's anxiety will be assessed using the modified Yale Preoperative Anxiety Scale-Short Version at the preoperative holding area before receiving medication (Time 1), and in the operating room after separation from the parent (Time 2).
     For each domain the patient's partial score will be divided by the maximum score obtainable in that domain (6 for the vocalizations domain and 4 for the remaining). The produced values for each domain are all added up and multiplied by 25. A score ranging from 22.92 to 100 will be obtained with higher values, representing higher states of anxiety. Thus, children with scores more than 30 will be considered as having anxiety and children with scores from 22,92 to 30 will be considered as not having experienced significant anxiety.
  2. Degree and onset of sedation will be assessed 15 and 30 minutes after administration of premedication by Ramsay sedation scale. Scale scored from 1 (least sedated) to 6 (most sedated).
acceptance of premedication | after ingestion of the premedication and before the surgery starts
  on a three-point scale. The score of 1 and 2 will be considered as satisfactory mask acceptance. The score of 3 and 4 will be considered as satisfactory mask acceptance.
  1. = Excellent (unafraid, cooperative, and accepts mask easily).
  2. = Good (slight fear of mask, easily reassured).
  3. = Fair (moderate fear of mask, not calmed with reassurance).
  4. = Poor (terrified, crying, or combative).
Time to recovery | immediately after the surgery average 2 hours postoperative
  1. Emergence time (minutes): from discontinuation of anaesthesia to opening eyes spontaneously
  2. Recovery time (minutes): from discontinuation of anaesthesia to a score of 8 on the modified Aldrete score

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed S. Shehab, Principal Investigator — Alexandria University
Locations (1):
- Ahmed S. Shehab, Alexandria, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
there is a plan to make individual participant data (IPD) collected in this study, including data dictionaries, available to other researchers
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After study ends upon request
Access Criteria: Accessible through the web site

REFERENCES:
- [Background] Bergendahl H, Lonnqvist PA, Eksborg S. Clonidine in paediatric anaesthesia: review of the literature and comparison with benzodiazepines for premedication. Acta Anaesthesiol Scand. 2006 Feb;50(2):135-43. doi: 10.1111/j.1399-6576.2006.00940.x. PMID 16430532
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/16430532/